CLINICAL TRIAL: NCT03977623
Title: Prospective Cohort Study for Genomic Evaluation in Patients With Diffuse Large B Cell Lymphoma After First Relapse/Progression
Brief Title: Genomic Evaluation in Patients With Diffuse Large B Cell Lymphoma After First Relapse/Progression
Acronym: COGET-B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Principal Investigator, Samsung Medical Center
Other Study IDs: 2019-04-087
Record Dates: First submitted 2019-05-17; First posted 2019-06-06 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood sample : SST(Serum Separation Tube) 3ml, EDTA (Ethylenediaminetetraacetic Acid) 3ml
  2. Tissue : unstained slides ((at least) 5 slides with a thickness of 5 microns)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DLBCL has the highest frequency out of all lymphoid malignancies. With the recent development of antitumor agents targeting intracellular/extracellular cell signaling pathways, patients have access to various treatment options after relapse. Therefore, for the purpose of developing effective treatment strategies, large-scale genomic data accumulation is necessary to understand the mechanism of relapse and refractory state of DLBCL.

DETAILED DESCRIPTION:
* To understand the mechanism of relapse by genome sequencing with tissues/blood obtained at diagnosis and relapse in patients with diffuse B cell lymphoma who relapsed after standard chemotherapy, to evaluate their response and survival following a salvage therapy depending on the genomic sequencing results, and to understand the prognostic or predictive value of genomic mutation.
* To understand the predictive value of genetic information with regard to the response to salvage chemotherapy and survival outcome in patients with newly diagnosed/relapsed or refractory large B cell lymphoma
* To determine the association between gene mutation, treatment response and prognosis in relapsed/refractory diffuse large B cell lymphoma (DLBCL), and to develop a clinically applicable platform by establishing a genetic data register based on prospective studies

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed DLBCL
* DLBCL who relapsed or were refractory to first-line treatment with rituximab-based immunotherapy
* Available for genomic analysis of tissues both at diagnosis (paraffin-embedded and stored) and at relapse (paraffin-embedded)
* Aged ≥18 years
* Written informed consent for participation in the prospective cohort study
* Written informed consent to peripheral blood collection and genetic testing of human tissues

Exclusion Criteria:

* No lymphoid malignancy, e.g. myeloid leukemia
* Any of the following lymphoid malignancies:

  1. Plasma cell dyscrasia, amyloidosis
  2. Hodgkin lymphoma
  3. Subtypes of B cell non-Hodgkin lymphoma, other than DLBCL
  4. T or NK(Natural Killer) cell non-Hodgkin lymphoma
  5. Other diseases in the WHO(World Health Organization) classification of lymphoid malignancies
* Experienced a relapse before
* Insufficient or no tissue sample at diagnosis for genomic analysis
* Can not understand or provide written informed consent
* Who do not provide written informed consent to blood collection and genetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects-both inpatients and outpatients-will be given an explanation of the significance of this study before recruitment.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Next generation sequencing with tumor tissue | 2-year follow-up from the end of the enrollment
  To understand the mechanism of relapse, targeted sequencing based on HemaScan panel including the essential genes (including 425 whole exome).
Next generation sequencing with blood | 2-year follow-up from the end of the enrollment
  To understand the mechanism of relapse, targeted sequencing based on HemaScan panel including the essential genes (including 425 whole exome).

SECONDARY OUTCOMES:
Data which included salvage chemotherapy. | 2-year follow-up from the end of the enrollment
  Progression free survival, response rate for salvage chemotherapy.
Data which included survival outcome. | 2-year follow-up from the end of the enrollment
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
* Data management of this clinical trial should be done in accordance with the ICH(International Conference on Harmonization)-GCP(Good Clinical Practice) and KGCP (Korean Good Clinical Practice)guidelines. To ensure the anonymity of subjects, each subject will be identified and managed by a randomly assigned subject number, instead of his/her name, in all documents so that persons not involved in the study could not identify subjects from their personal data.
  * Subjects participating in this clinical trial may have to provide some of their personal information, but such information will not be directly used or necessary in the study but will be used only for the purpose of connecting clinical data obtained for the clinical trial. Collected information will be used until the clinical trial report is complete.